CLINICAL TRIAL: NCT02991573
Title: Clinical Post-Market Surveillance Study of Ceram.x Universal and Prime&Bond Universal When Used for Class II Restorations at the University of Sheffield
Brief Title: Clinical Study Class II on Ceram.x Universal and Prime&Bond
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STH18842 CIP 14.1515
Record Dates: First submitted 2015-12-04; First posted 2016-12-13 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2019-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- existing adhesive (control) (Active Comparator): control adhesive
  Interventions: Device: Ceram X; Device: Prime & Bond XP
- new adhesive: technique 1 (Experimental): Prime & Bond Universal: technique 1
  Interventions: Device: Prime & Bond Universal; Device: Ceram X; Procedure: technique 1
- new adhesive: technique 2 (Experimental): Prime & Bond Universal: technique 2
  Interventions: Device: Prime & Bond Universal; Device: Ceram X; Procedure: technique 2

INTERVENTIONS:
Device: Prime & Bond Universal — Prime & Bond Universal
  Arms: new adhesive: technique 1; new adhesive: technique 2
Device: Ceram X
Device: Prime & Bond XP — Control
  Arms: existing adhesive (control)
Procedure: technique 1
  Arms: new adhesive: technique 1
Procedure: technique 2
  Arms: new adhesive: technique 2

SUMMARY:
Damage to teeth from decay or previous old silver fillings can be repaired with tooth-coloured filling materials that stick to the tooth. These materials have been around for some years and have become more sophisticated; with greater ease of placement by the dentist and better durability for the patient. The fillings are designed to be used in combination with a specific glue (adhesive) that is designed to stick to the different parts of the tooth to provide a good seal, the outer enamel and the inner dentine.

This study will examine the performance of a state-of-the-art modern tooth coloured filling material (Ceram X) in combination with an existing adhesive (control adhesive) and a new adhesive (Prime & Bond Universal) used in two different techniques; both of which are known to work but one is easier to apply. This results in three treatment groups.

At the start of the study, the test material Prime&Bond Universal is CE-marked, as are all other medical devices used. Thus, this study is not conducted to meet any regulatory requirements. The rationale of this study is the extension of knowledge primarily concerning the clinical performance of Prime&Bond Universal in molars.

Two investigators (to be confirmed) will place a minimum of 25 restorations per group (75 restorations in total) to assess the performance of the materials in a comparative design. The study restorations will be monitored for a period of 18 months (with the option to extend the evaluation period to 48 months).

After placement of restorations under controlled clinical conditions, the primary objective of the study is the determination of post-operative sensitivity and pulp vitality, marginal adaptation and staining of margins of the restorations. In addition, fracture of material and retention, recurrent caries, occlusal contour and wear, approximal anatomical form will be determined as well as the failure rate as defined by the ADA.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patient selection:

* Patients of either gender and at least 18 years old at the start of the study (enrollment), who are seeking treatment at the dental clinic involved, will be invited to participate in the study if they are in need of at least one eligible Class II posterior restoration in a permanent molar.

Tooth inclusion criteria:

* Per patient, a maximum of three Class II restorations will be included. If three restorations are indicated and eligible, one of each material will be included.
* Vital, non-symptomatic permanent teeth with Class II lesions are suitable for inclusion into the study if the following criteria are met:

  * - location: first or second molars (ADA guidelines[1]);
  * - restoration size: moderate: no cusp replacements;
  * - cavity size: occlusal width ≥ 1/3 of intercuspal distance (ADA guidelines[1]);
  * - cavity outline: preparation to include a proximal box with or without an occlusal step;
  * - box: cervical outline in enamel;
  * - occlusion: at least one opposing contact point in enamel.
* Enrollment of patients will continue until the specified minimum number of restorations per group (N=25) and/or the minimum number of patients (N=50) have been reached.

Exclusion Criteria:

Exclusion criteria for patient selection:

* The exclusion criteria (i.e. contraindications) as described in the Instructions for Use of the test, control and restorative materials apply:
* Use with patients who have a history of severe allergic reaction methacrylate resins or any of the components; direct application to dental pulp (direct pulp capping).
* Patients who are unable to give informed consent or vulnerable population as defined in ISO 14155[4] will not be enrolled.

Tooth exclusion criteria:

As a rule, the materials are not to be used in situations as specified in the Instructions for Use - Section Contraindications.

* direct or indirect pulp-capping Furthermore, teeth with class II lesions are excluded when involved with
* inflammation or pulpitis (pain),
* periodontitis with probing depth > 6 mm,
* extraction of tooth to be expected within the next 12 months,
* signs of strong parafunctions or erosion (exposed dentin on occlusal surface and/or wear facets > 6 mm2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related postoperative sensitivity recorded as a change from baseline to that reported at 14 days, 6 months, 12 months and 48 months, assessed using a visual analog scale. | 14 days, 6 months, 12 months and 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martin, Professor, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Professor Nicolas Martin, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No